CLINICAL TRIAL: NCT03930290
Title: Vaginal Tactile Imaging for the Assessment of Physiologic Elasticity Changes During Pregnancy and After Labor.
Brief Title: Physiologic Elasticity Changes During Pregnancy and After Labor.
Status: Terminated | Type: Observational
Why Stopped: Difficulty in patient recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal Investigator, Rambam Health Care Campus
Other Study IDs: 0567-18-RMB
Record Dates: First submitted 2019-04-25; First posted 2019-04-29 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Vaginal Prolapse
MeSH Terms: conditions — Uterine Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant patients: Pregnant patients in their 2nd trimester.
  Interventions: Diagnostic Test: Vaginal tactile imager

INTERVENTIONS:
Diagnostic Test: Vaginal tactile imager — Vaginal elasticity evaluation by vaginal tactile imaging analysis.

SUMMARY:
Female pregnant patients in their 2nd trimester will be evaluated for vaginal elasticity using vaginal tactile imaging in addition to elasticity evaluation during the 3rd trimester and 6 weeks postpartum.

DETAILED DESCRIPTION:
Female pregnant patients in their 2nd trimester will be evaluated for vaginal elasticity using vaginal tactile imaging. Vaginal elasticity will also be evaluated during the 3rd trimester and 6 weeks postpartum.

Patients will be recruited and sign a consent form. Assessment of vaginal elasticity via vaginal tactile imaging will be performed at 3 different points:

* During the 2nd trimester.
* During the 3rd trimester.
* 6 weeks postpartum. Every patient will serve as her own control. Demographic, gynecologic and obstetric history will be obtained from patients' electronic files.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients in their 2nd trimester.

Exclusion Criteria:

* Pregnant patients presenting after their 2nd trimester.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnancy
Study Population: Pregnant patients in their 2nd trimester with no regard to previous obstetric history.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Vaginal elasticity | From the beginning of the 2nd trimester of pregnancy up to 6 weeks postpartum.
  Vaginal elasticity evaluation by vaginal tactile imaging analysis

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam healthcare campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided